CLINICAL TRIAL: NCT01317810
Title: A Phase 4, Observational, Non-interventional Study Measuring and Tracking Changes in Overactive Bladder Medication and/or Overactive Bladder Medication Dose in Subjects With Overactive Bladder
Brief Title: A Study Measuring and Tracking Changes in Overactive Bladder (OAB) Medication
Status: Withdrawn | Type: Observational
Why Stopped: Corporate decision not to initiate the trial
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Clinical Trials Registry, Astellas Pharma US, Inc
Other Study IDs: 905-UC-060
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Overactive Bladder (OAB)
Keywords: Overactive Bladder (OAB); Observational; Registry
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Overactive Bladder (OAB): Combination of new OAB subjects and existing subjects on OAB medication

SUMMARY:
The purpose of this study is to track changes in overactive bladder (OAB) medical regimen and/or OAB medication dosage requirements.

DETAILED DESCRIPTION:
Subjects will complete a study specific survey questionnaire at Screening and the Month 1 through Month 6 visits. Subjects will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has overactive bladder as determined by their prescribing physician
* Subject is currently receiving pharmacotherapy for overactive bladder
* Subject is willing to comply with required protocol/study requirements

Exclusion Criteria:

* Subject has a history of a clinically significant illness or medical condition prior to screening that would preclude participation in the study
* Male subjects with Lower Urinary Tract Symptoms (LUTS) or Bladder Outlet Obstruction (BOO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with overactive bladder (OAB)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in overactive bladder (OAB) medication/ treatment regimen | 6 months
Reason for change in OAB medication/treatment regimen | 6 months

SECONDARY OUTCOMES:
Persistence of use of any OAB medication as reported by the Physician | 6 months
Change in OAB medication including discontinuation of OAB medication as reported by the Physician | 6 months
Subject reported efficacy | 6 months
  Measured by the Subject Survey Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development, Inc.